CLINICAL TRIAL: NCT05923749
Title: A Prospective Randomised Controlled Study Demonstrating the Clinical Benefit of Biatain® Ag Relative to Cutimed® Siltec® Sorbact® for the Treatment of Venous Leg Ulcers
Brief Title: A RCT Evaluating the Clinical Benefit of a Silver Dressing in the Treatment of Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP354
Record Dates: First submitted 2023-06-14; First posted 2023-06-28 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Wound Heal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Biatain Ag (Experimental)
  Interventions: Device: Biatain Ag
- Cutimed Siltec Sorbact (Active Comparator)
  Interventions: Device: Cutimed Siltec Sorbact

INTERVENTIONS:
Device: Biatain Ag — Biatain with silver
  Arms: Biatain Ag
Device: Cutimed Siltec Sorbact — comparator device
  Arms: Cutimed Siltec Sorbact

SUMMARY:
Approximately 178 patients with a venous leg ulcer will be included in the investigation evaluating wound healing. All subjects are randomized to one of two treatment arms with an intervention period of 4 weeks followed by a 8 week standard of care period.

ELIGIBILITY:
Inclusion Criteria:

* Has signed informed consent
* Is above 18 years of age or above and has full legal capacity
* Has venous leg ulcer (C6 of the CEAP classification) with a duration longer than 4 weeks but no longer than 5 years
* Has acceptance of compression bandages
* Has a wound at risk of infection based on WAR (wounds at risk of infection) score with score of ≥3 points OR has at least three of the following clinical signs of bacterial contamination based on the Therapeutic index for local infections (TILI) score:

  * Erythema to surrounding skin
  * Heat
  * Oedema, induration or swelling
  * Spontaneous pain or pressure pain
  * Stalled wound healing
  * Increase and/or change of color or smell of exudate
* Has wound area of min 1x1 cm and max 10x10 cm
* Has wound with depth of max 2 cm
* Has wound with medium to high level of exudate (but should not require more than 1 dressing change/day)
* Has ankle-brachial pressure (ABI) ≥0.8 AND, for patients with diabetes mellitus, additional biphasic Doppler signal up to the ankle
* Ability (assessed by the investigator) and willingness to adhere to a 1-month intervention period
* For patients with diabetes, has HbA1c ≤ 10%/≤ 86 mmol/mol, measured within the last 3 months prior to inclusion
* Should be able to follow the study protocol with the prescribed cleansing product (NaCl) and dressing

Exclusion Criteria:

* Is pregnant or breastfeeding
* Has wounds with exposed tendons, bones, fistulas. Or wounds with cavity, undermined or tunnelling
* Has infection requiring antibiotics (also for other reasons than wound infection) OR has received antibiotics within the last 1 week before inclusion
* Has been receiving the following medical treatment within the last 4 weeks: immunosup-pression, immunomodulating, cytostatic medi-cation or corticoids (topical except for in the wound, inhalation, and stable systemic treat-ment up to 5 mg per day (stable defined as minimum 4 weeks) is allowed
* Has a systemic hematological disease
* Has renal insufficiency requiring dialysis
* Has advanced heart failure NYHA III/IV
* Has a psychiatric illness that inhibits compliance with the study protocol
* Has severe congenital immunodeficiency such agammaglobulinemia, severe combined immunodeficiency (SCID)
* Has allergy towards silver or other dressing ingredients (including compression therapy)
* Has wound with > 50% necrotic tissue
* Treatment of wound with an anti-microbial wound dressing within the last 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Wound healing | After 4 weeks
  Relative wound area change measured by calculation of area based on photo of wound

SECONDARY OUTCOMES:
Wound area reduction | After 4 weeks
  Reaching ≥ 40% wound area change
Wound healing | After 12 weeks
  Wounds healed after 12 weeks (yes/no assessed by investigator)
Quality of Life (based on Wound-Quality of Life-17 questionnaire) | After 4 and 12 weeks
  Patient Quality of Life

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - Royal Research, Corp., Hollywood, Florida
  - Three Rivers Wound and Research Center, North Port, Florida
  - Detroit foot and ankle Specialists, Clinton Township, Michigan
  - SerenaGroup Research Center Omaha, Omaha, Nebraska
  - Serena Group, Monroeville, Pennsylvania
- Dermato-Venerologisk Afd, Copenhagen, Denmark
- Germany (6):
  - Wundmanagement Gefäßzentrum Aachen Wundmanagement, Aachen
  - Katholisches Klinikum Bochum, Bochum
  - Krankenhaus Buchholz und Winsen gemeinnüzige GmbH, Buchholz
  - ProDerma, Dülmen
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Giessen und Marburg GmbH, Giessen
- Pioneer Wound Healing and Lymphedema centres, Eastbourne, United Kingdom

IPD SHARING:
Plan to Share IPD: No